CLINICAL TRIAL: NCT04946396
Title: Evaluation of the Effects of Continuous Dexmedetomidine Infusion on Systemic Microvascular Function in Patients Undergoing Laparoscopic Cholecystecthomy: a Prospective Study
Brief Title: Effects of Continuous Dexmedetomidine Infusion on Systemic Microvascular Function in Laparoscopic Cholecystecthomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 47593521.1.0000.5279
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Surgery
Keywords: dexmedetomidine; microcirculation; general anesthesia; central alpha-2 agonists; tissue perfusion
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups of 35 patients each: 1) patients who will receive continuous intraoperative infusion of dexmedetomidine hydrochloride (0.5 µg/kg/h) (DEX group) or 2) control group, patients who will receive continuous infusion of 0.9% saline solution (CONT group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine intravenous infusion (Experimental): Patients who will receive continuous intraoperative infusion of dexmedetomidine hydrochloride (0.5 µg/kg/h).
  Interventions: Drug: dexmedetomidine intravenous infusion
- 0.9% saline solution intravenous infusion (Sham Comparator): Patients who will receive continuous infusion of 0.9% saline solution (sham group).
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: dexmedetomidine intravenous infusion — Dexmedetomidine intravenous infusion during laparoscopic cholecystecthomy
  Arms: dexmedetomidine intravenous infusion
Drug: 0.9%sodium chloride — 0.9%sodium chloride intravenous infusion during laparoscopic cholecystecthomy
  Arms: 0.9% saline solution intravenous infusion

SUMMARY:
The microcirculation represents the primary site of exchange of oxygen and nutrients for tissues, and the preservation of microcirculatory perfusion is essential for the maintenance of organ function. The microcirculation is extremely dynamic and may vary according to the individual's temperature, systemic blood pressure, the use of medications, during physical and mental activity, age and pathological processes. In this context, the development of portable microscopes for clinical use has made possible the non-invasive visualization of the microcirculation and tissue perfusion in patients undergoing several highly complex procedures in cardiology, including cardiac surgery with cardiopulmonary bypass, ECMO (Extracorporeal Membrane Oxygenation) and in critically ill patients in intensive care.

CytoCam, for example, is a handheld device that incorporates a darkfield incident light illumination system with a series of high-resolution lenses that project images to a computer dedicated to the system. Dexmedetomidine is a selective agonist of 2-adrenergic receptors in the central nervous system, whose administration results in a reduction in the activity of the sympathetic nervous system and a reduction in the systemic release of catecholamines. Its use in the perioperative period has several beneficial effects, such as reducing neuroendocrine and hemodynamic responses due to anesthesia and surgery, through induction of sedation and analgesia, in addition to reducing the consumption of opioids and anesthetics in general. Several recent studies report that the use of dexmedetomidine in the perioperative period reduces the incidence of postoperative complications, reduces the time on mechanical ventilation and attenuates the neuroendocrine response due to surgical trauma and extracorporeal circulation in patients undergoing cardiac surgery. However, the effects of dexmedetomidine on systemic microcirculation function during its use in anesthesia for elective surgical procedures of medium complexity are not yet known. In conclusion, the hypothesis of the present study is that continuous intravenous infusion of dexmedetomidine during balanced general anesthesia increases the microvascular perfusion flow rate in the sublingual mucosa, representing an increase in systemic microvascular perfusion.

DETAILED DESCRIPTION:
CytoCam, is a handheld device that incorporates a darkfield incident light illumination system with a series of high-resolution lenses that project images to a computer dedicated to the system. Dexmedetomidine is a selective agonist of 2-adrenergic receptors in the central nervous system, whose administration results in a reduction in the activity of the sympathetic nervous system and a reduction in the systemic release of catecholamines. Its use in the perioperative period has several beneficial effects, such as reducing neuroendocrine and hemodynamic responses due to anesthesia and surgery, through induction of sedation and analgesia, in addition to reducing the consumption of opioids and anesthetics in general. Several recent studies report that the use of dexmedetomidine in the perioperative period reduces the incidence of postoperative complications, reduces the time on mechanical ventilation and attenuates the neuroendocrine response due to surgical trauma and extracorporeal circulation in patients undergoing cardiac surgery. However, the effects of dexmedetomidine on systemic microcirculation function during its use in anesthesia for elective surgical procedures of medium complexity are not yet known. In conclusion, the hypothesis of the present study is that continuous intravenous infusion of dexmedetomidine during balanced general anesthesia increases the microvascular perfusion flow rate in the sublingual mucosa, representing an increase in systemic microvascular perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes (age ≥ 18 and ≤ 60 years)
* Physical state ASA I or II according to the criteria of the American Association of Anesthesiology
* Planned surgery of cholecystectomy by videolaparoscopy

Exclusion Criteria:

* Patient's refusal to participate in the study
* Inflammation or infection in the sublingual mucosa
* Emergency surgery
* Grade III obesity (BMI ≥39.9 kg/m2)
* Pregnancy or lactation
* Autoimmune diseases, malignant neoplasms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
change in microvascular flow index | during surgery
  sublingual microvascular density

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO TIBIRICA, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- Eduardo Tibiriçá, Rio de Janeiro, Brazil